CLINICAL TRIAL: NCT04960774
Title: Human Subject Research Ethics Committee, 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Brief Title: Risk Factors for Severe Periodontitis in 30 to 40 Year Olds: a Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0184
Record Dates: First submitted 2021-06-16; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-04

CONDITIONS: Severe Periodontitis; Risk Factors; Gene Polymorphism
MeSH Terms: conditions — Periodontitis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients with non-severe periodontitis or healthy people who were treated in our department in the same period were included as the control group.
  Interventions: Other: Observational study, no intervention
- Severe periodontitis group: Severe periodontitis patients who meet the inclusion and exclusion criteria in the Department of Stomatology, the second affiliated Hospital of Medical College of Zhejiang University
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention — Observational study, no intervention

SUMMARY:
Periodontitis is one of the most common oral diseases, which is characterized by alveolar bone resorption and destruction. In China, as a major country in the incidence of periodontitis, there is a huge population of patients with severe periodontitis, and the incidence rate is as high as 12.1-16.1% . Previous studies have suggested that the prevalence and severity of periodontal disease increase with age. However, recent articles on meta analysis and related epidemiological investigations suggest that the prevalence of severe periodontitis does not increase with age, and the prevalence of SP remains at about 10% even in the elderly. In order to comprehensively analyze the risk factors of this population, it is inseparable from the analysis of gene polymorphism. At present, it is considered that the main genes that may be related to the severity of periodontitis are IL-1 α-889, rhIL-talk 1 β + 3953, 6-174, 10-597, CD14-260, CD14-159, MMP1-1607 and so on, which may be related to the severity of periodontitis.

DETAILED DESCRIPTION:
Periodontitis is one of the most common oral diseases, which is characterized by alveolar bone resorption and destruction. In 2010, severe periodontitis (severe periodontitis,SP) had become the sixth largest epidemic disease in the world, affecting 10.8% of the global population or 743 million people . In China, as a major country in the incidence of periodontitis, there is a huge population of patients with severe periodontitis, and the incidence rate is as high as 12.1-16.1% . The fourth National Oral Health Epidemiological Survey also found that the oral health of residents aged 35-44 is generally poor , which has become a major obstacle to the implementation of the "Healthy China 2030" strategy. Previous studies have suggested that the prevalence and severity of periodontal disease increase with age . The possible reasons for this phenomenon are as follows.First, the cumulative effect of attachment level and bone loss with age.Second, changes related to the aging process, such as drug intake, decreased immune function, and changes in nutritional status interact with risk factors can increase the susceptibility to periodontitis. However, recent articles on meta analysis and related epidemiological investigations suggest that the prevalence of severe periodontitis does not increase with age, and the prevalence of SP remains at about 10% even in the elderly. In addition, the global meta analysis with large sample size showed that the prevalence of SP increased sharply between 30 and 40 years old, peaked at about 38 years old. This trend of severe periodontitis with age is not consistent with our traditional cognition, and there is no related research to explain this trend. However, it is found that 30-40 years old patients with severe periodontitis account for a large proportion, so it is of great significance to analyze the risk factors of this group and carry out targeted prevention and control. In order to comprehensively analyze the risk factors of this population, it is inseparable from the analysis of gene polymorphism. Studies related to severe periodontitis gene polymorphism are mainly focused on Toll-like receptor (Toll-likereceptors), interleukin (interleukin,IL), immunoglobulin receptor (Immunoglobulinreceptors), formyl peptide receptor (Formylpeptide receptor), vitamin D receptor (VitaminDreceptor, VDR) and matrix metalloproteinases (matrixmetalloproteinase,MMP). At present, it is considered that the main genes that may be related to the severity of periodontitis are IL-1 α-889, rhIL-talk 1 β + 3953, 6-174, 10-597, CD14-260, CD14-159, MMP1-1607 and so on, which may be related to the severity of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patients aged between 30 and 40 years old were diagnosed with severe periodontitis and were treated for the first time, while those in the control group were patients with non-severe periodontitis or healthy people. All the subjects had complete basic information, questionnaire data and clinical examination data. 3. The patient's thinking is clear, there is no barrier to communication, and can cooperate to complete the questionnaire. 4.In addition, the genetic polymorphism test required that the three generations were all Han nationality, with no history of orthodontic treatment, no obvious malocclusion and local stimulating factors, and no Systemic disease (including diabetes, cardiovascular disease, hepatitis, HIV infection, etc.), non-smoking or non-smoking for more than 5 years

Exclusion Criteria:

* 1. Patients suspected to be invasive periodontitis, the plaque level and the degree of periodontal destruction are disproportionate. 2. Systemic diseases (including diabetes, cardiovascular disease, hepatitis, HIV infection, etc.) 3. Pregnant women, women who are pregnant, lactating or mentally ill. 4.Those who are taking known drugs that affect periodontal tissue or have a history of antibacterial treatment within 6 months. 5.Those who have a history of periodontal treatment within 6 months are excluded. 6.In addition, testing for genetic polymorphism required the exclusion of malignancies or those who had undergone radiotherapy or chemotherapy

Ages: 30 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: According to the CDC/AAP case definition (Page&Eke2007/Page&Eke2012) 1. No periodontitis is defined as no indication of mild, moderate or severe periodontitis; 2. Mild periodontitis is defined as the loss of attachment level at the adjacent site of ≥ 2 teeth ≥ 3mm and the periodontal probing depth ≥ 4mm (not on the same tooth) at the adjacent site of ≥ 2 teeth or having a site periodontal probing depth ≥ 5mm. Moderate periodontitis is defined as the loss of attachment level ≥ 4mm (not on the same tooth) at the adjacent site of ≥ 2 teeth, or periodontal probing depth ≥ 5mm (not on the same tooth) at the adjacent site of ≥ 2 teeth. Severe periodontitis is defined as the loss of attachment level at the adjacent site of ≥ 2 teeth ≥ 6mm (not on the same tooth) and the periodontal probing depth ≥ 5 mm for the adjacent site of ≥ 1 tooth position. The third molar is not included.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
probing depth (PD) | For risk factor analysis, only the baseline is measured, which refers to the first visit
  The distance from the bottom of the periodontal pocket to the gingival margin (mm) was measured with a periodontal probe (UNC-15, Hu-Friedy, Chicago) parallel to the long axis of teeth. 6 sites including mesial, median and distal on the lips (cheek) and tongue surfaces were recorded for each tooth.
clinical attachment level (CAL) | baseline
  The distance from the gingival crevicular floor or periodontal pocket floor to the enamel bone boundary was measured by periodontal probe. The mesial, median and distal sites of the labial (buccal) surface and tongue surface of each tooth were measured.
Number of missing teeth | baseline
  Refers to the number of missing teeth except the third molar
  Refers to the number of missing teeth except the third molar
  Refers to the number of missing teeth except the third molar
  Refers to the number of missing teeth except the third molar
debris index (DI-S) | baseline
  The oral cavity was divided into 6 segments, and the debris of 6 index teeth was examined: 16, 26, 36, 46, 11, 31; if missing, check the adjacent teeth in the same area. The values are as follows: 0 = there is no debris on the tooth surface; 1 = the debris coverage area is less than 1/3; 2 = the debris coverage area is between 1/3 and 2/3; 3 = the debris coverage area accounts for more than 2/3 of the tooth surface.
calculus (CI-S) | baseline
  The examination method is the same as above, check the calculus condition of 6 index teeth. The assigned values are as follows: 0 = no supragingival and subgingival calculus; 1 = the area covered by supragingival calculus is less than 1 / 3 of the tooth surface; 2 = the area covered by supragingival calculus is between 1 / 3 and 2 / 3, or there are scattered subgingival calculi in the neck; 3 = the area covered by supragingival calculus accounts for more than 2 / 3 of the tooth surface, or there are continuous and thick subgingival calculus in the neck.
simplified oral hygiene index (OHI-S) | baseline
  The sum of the 6 CI-S or DI-S, choose the larger one. 0HI-S ≥ 10 means poor oral hygiene. OHI < 10 is good for oral hygiene.
Number of defective restorations | baseline
  It means that the crown edge of the restoration is located under the gingiva, the surface of the restoration is rough, the degree of fit with the tooth surface is not good, the shape is too convex, the contact area, marginal ridge recovery is not good, and so on. Among them, the fixed bridge is calculated according to the number of teeth of the bad bridge.
Gingival biotype | baseline
  According to the judgment method proposed by Kan et al, and combined with the clinical practice of our country, the periodontal biotypes are divided into the following three types: 1. Thick gingiva:. Examination methods: the outline of the periodontal probe into the gingival sulcus is completely unrecognizable at the gingival margin and through the gingival tissue at the front of the probe; 2. Thin gingiva: Examination method: the outline of the periodontal probe into the gingival sulcus can be recognized at the gingival margin and through the gingival tissue at the front of the probe . 3. Intermediate gingiva: the characteristic is between the above two; examination method: the outline of the periodontal probe into the gingival sulcus can be identified at the gingival margin through the gingival tissue, while the front part of the probe cannot be identified.
Dentition crowding degree | baseline
  The crowding degree of the canine-canine area of the lower anterior teeth can be easily evaluated according to the crowding degree of the canine-canine area of the lower anterior teeth, which can be divided into the following four grades : 0 = none, 1 = the crowding degree of the lower anterior teeth is equal to half the width of the lower central incisor, 2 = the crowding degree of the lower anterior teeth is equal to the width of a central incisor, 3 = the crowding degree of the lower anterior teeth exceeds the width
Molar relationship | baseline
  Angle class I: the occlusion of the mesiobuccal tip of the maxillary first molar is neutral with the molar in the mesiobuccal groove of the mandibular first permanent molar; Angle II: the distance of the mandibular retreating 4 molars or half of the premolars, the distance of the molars is distal; Angle III: the distance of the mandibular forward movement of at least 1x4 molars or half of the premolars, and the molars are mesial.
overjet | baseline
  The horizontal distance from the incisor edge of the upper incisor to the labial surface of the lower incisor. The distance within 3mm is normal coverage, 3mm < coverage ≤ 5mm is I-degree deep coverage, 5mm < coverage ≤ 8mm is II-degree deep coverage, and coverage > 8mm is III-degree deep coverage
overbite | baseline
  The front teeth cover the front teeth covering no super cut 1/3 and the lower teeth cutting in front of the front terture tongue is 1/3, and it is normal to cover it; I degree deep cover: up to teeth cover The lower teeth are more than 1/3 and less than 1/2 or lower tooth dumps are biting in front tootooth, and less than 1/3 and less than 1/2; II degree deep cover: up to teeth Over the previous lip surface exceeds the cut 1/2 and less than 2/3 or the until the until the front teeth are above the front tootooth tongue, the tongue is less than 2/3; III degree deep cover: upper teeth Override overhead lip surfaces exceed 2/3 or lower teeth in the front tooth tongue more than 1/3;
gender | baseline
  Divided into male and female
Nation | baseline
  It is divided into Han and non-Han
BMI | baseline
  Body mass index ((BMI)) = weight (kg) / height (m) squared according to the guidelines for the Prevention of overweight and Obesity in Chinese Adults [1]: BMI < 18.5 kg/m2 is weight loss 18.5 kg/ m2 < 24.0 kg/m2 is normal 24.0 kg/ m2 < 28.0 kg/m2 is overweight BMI ≥ 28.0 kg/m2 is obese
Educational level | baseline
  Senior high school ,below junior college ,undergraduate and above
Economic level | baseline
  The measure of economic level is reflected by the per capita monthly income of the family = the total monthly income of the family / the number of people in the family.
Mental stress | baseline
  Mental stress is measured by Perceptual Stress Scale.The scale makes necessary changes to the overall structure and specific items of PSS to make the content more in line with China's national conditions. CPSS consists of 14 items, which are composed of two dimensions: the sense of tension and the sense of loss of control. Using Likert's five-point scoring system, 1 means "never", 2 means "occasionally", 3 means "sometimes", 4 means "often" and 5 means "always". The total score of the scale ranges from 14 to 70, and the higher the score, the greater the perceived pressure.
Smoking | baseline
  Smoking status is constructed by two questions in the questionnaire: subjects who smoke every day or a few days and smoke more than 100 cigarettes; former smokers: subjects who do not smoke at present but have smoked more than 100 cigarettes in the past; non-smokers: subjects who smoked no more than 100 cigarettes.
History of orthodontic treatment | baseline
  Past history of orthodontic treatment , during orthodontic treatment ,no orthodontic treatment
Food impaction history | baseline
  Number of food impactions in the past 6 months
Bruxism / clenched teeth | baseline
  Whether others tell or feel that they are grinding and / or clenching their teeth during sleep; or whether there is unconscious clenching and / or grinding during the day
Unilateral mastication habit | baseline
  Had the habit of chewing on one side in the past
Last Dental Visit | baseline
  Includes all professional stomatologists, not just periodontists.
Oral health care self-efficacy | baseline
  Oral health self-efficacy was evaluated by Wu Di's Chinese oral health self-efficacy scale.A total of 15 items in this scale are divided into 3 dimensions, namely, oral self-efficacy, correct tooth brushing self-efficacy and balance, diet self-efficacy. Using the likert5 score scale, the score was from 1 (no confidence at all) to 5 (very confident). The total score was 15-75, in which the score was 15-53 as low performance, 54-59 as medium performance, and 60-75 as high performance. The higher the score, the higher the level of oral health self-efficacy.
Tooth brushing | baseline
  mode, frequency, time of Tooth brushing
auxiliary equipment using | baseline
  The use of other auxiliary equipment such as dental floss.Including tooth brush, tooth punch, etc., but excluding toothpicks and mouthwash
Regular scaling | baseline
  the habit of cleaning teeth regularly for half a year to one year
Genotypic polymorphism | baseline
  allele frequency of IL-1α-889，IL-1β
  +3953，IL-6-174，IL-10-597，CD14-260，CD14-159，MMP1-1607

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Lihong, Hangzhou, China